CLINICAL TRIAL: NCT00794092
Title: Magnetic Resonance Imaging of Aortic Aneurysm Instability
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007/R/CAR/15
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sinerem (Experimental): MRI scanning of patients with AAA before and 24hrs +/- 4hrs after administration of Sinerem
  Interventions: Drug: Sinerem administration

INTERVENTIONS:
Drug: Sinerem administration — Single dose

SUMMARY:
Abdominal aortic aneurysm (AAA) is a progressive enlargement of the aorta, the largest blood vessel in the body. It is at risk of bursting when it is usually fatal. Currently the risk of the AAA bursting is estimated from its diameter. In this study, the investigators hope to develop a new type of aneurysm scan involving Magnetic Resonance Imaging (MRI). It is hoped that this scan will be better at determining which AAAs are at risk of bursting and therefore require an operation to prevent this.

DETAILED DESCRIPTION:
Abdominal aortic aneurysms (AAA) have a prevalence of ~5% and when ruptured carry a mortality rate of ~90%. The pathophysiology of AAA encompasses a range of poorly understood biomechanical and biological processes. Currently the diameter of the aneurysm is used as a surrogate for the risk of rupture and patients with an aneurysm diameter greater than 55 mm are considered for elective surgical repair. However, this reliance on a single surrogate measure is too simplistic and does not take into account other physical and biological aspects of the AAA. We propose to evaluate the role of inflammation, proteolysis and neovascularisation in patients with AAA disease. We will compare novel magnetic resonance imaging techniques with blood and tissue measures of inflammation (c-reactive protein, cytokines, macrophage and leucocyte density), proteolytic activity (matrix metalloproteinases, tissue inhibitors of metalloproteinases) and neovascularisation (vessel density, endothelial progenitor cells). By comparing findings between patients with symptomatic and asymptomatic disease, this study will inform our understanding of the disease process as well as potentially identify risk markers of AAA instability that could be used to follow-up patients with asymptomatic disease.

ELIGIBILITY:
Inclusion Criteria:

* AAA measuring >40mm in AP diameter on ultrasound scanning
* Age >40 years (patients younger than this with AAA may have a connective tissue disorder and a different aetiology to their disease)
* Considered to be suitable for standard infra-renal open surgical repair

Exclusion Criteria:

* Patients who are not deemed to be fit for open surgical repair
* Patients who are deemed to be suitable for a stent graft performed by the radiologists rather than the standard operation
* Contraindication to MRI scanning identified from MRI Safety Questionnaire (see attached)or claustrophobia
* Age <40 years
* Patients requiring emergent repair such that there is insufficient time available to complete the protocol
* Patients refusing to give consent
* Patients unable to give consent
* Pregnant women (contrast is teratogenic in animals)
* Intercurrent illness (may confound the results)
* Patients with a systemic inflammatory disorder or underlying malignancy
* Patients who require an emergency operation such that there is insufficient time to complete the study protocol
* Renal dysfunction (Creat >250 or eGFR<25)
* Hepatic dysfunction (Child's grade B or C)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change in signal intensity in a Region of Interest on MRI scanning | 24 hours after administration of Sinerem

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh/Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom

REFERENCES:
- [Result] Richards JM, Semple SI, MacGillivray TJ, Gray C, Langrish JP, Williams M, Dweck M, Wallace W, McKillop G, Chalmers RT, Garden OJ, Newby DE. Abdominal aortic aneurysm growth predicted by uptake of ultrasmall superparamagnetic particles of iron oxide: a pilot study. Circ Cardiovasc Imaging. 2011 May;4(3):274-81. doi: 10.1161/CIRCIMAGING.110.959866. Epub 2011 Feb 8. PMID 21304070